CLINICAL TRIAL: NCT04125914
Title: HEALTH4Families: Optimizing a Weight Management and Health Behavior Intervention for BRCA+ and Lynch Syndrome Families
Brief Title: Weight Management and Health Behavior Intervention in Lowering Cancer Risk for BRCA Positive and Lynch Syndrome Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0775; NCI-2019-02453 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0775 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-05-06; First posted 2019-10-14 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hereditary Breast Carcinoma; Hereditary Ovarian Carcinoma; Lynch Syndrome
MeSH Terms: conditions — Breast Cancer, Familial; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Health Promotion; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (weight management, health behavior intervention) (Experimental): Participants undergo weight management and health behavior intervention with a combination of 4 components for 16 weeks. TELEPHONE COACHING: Participants receive 1 phone call each week from a coach over 30-45 minutes to discuss diet, physical activity and goal setting. EMAIL COACHING: Participants receive 1 phone call to discuss the process over 10-15 minutes and then receive 1 email each week for 16 weeks. NO COACHING: Participants receive 1 phone call the first week over 10-15 minutes to discuss the process. TEXT MESSAGING: Participants receive 7-12 text messages comprising information about diet and physical activity each week for 16 weeks. SELF-MONITORING: Participants record their food intake and weight directly into the Fitbit website or application 4-7 days each week or 1 day each week for 16 weeks. FAMILY TEAM INTERVENTION: Participants receive 2 group phone calls and join a Facebook group that is monitored by research staff where they can interact with each other and coaches.
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: E-mail; Behavioral: Exercise Intervention; Other: Health Promotion and Education; Other: Internet-Based Intervention; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Record food intake
Other: E-mail — Receive e-mails
  Other Names: Electronic Mail; Email
Behavioral: Exercise Intervention — Undergo exercise
Other: Health Promotion and Education — Receive text messages
Other: Internet-Based Intervention — Join Facebook page
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive telephone coaching

SUMMARY:
This trial studies how well weight management and health behavior intervention works in helping patients with hereditary breast and ovarian cancer and Lynch syndrome mutation carriers lose or maintain a healthy weight and lower their risk for cancer. Lifestyle behaviors such as physical activity, diet, and weight management may play a key role in preventing cancers and improving outcomes even in those with hereditary cancer syndromes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify the most effective intervention components for weight loss (primary outcome) and percent energy from fat, vegetable and fruit consumption, physical activity, and theory based behavioral determinants (secondary outcomes), with the goal of developing an optimized weight management intervention for hereditary breast and ovarian cancer (HBOC) and Lynch syndrome (LS) mutation carriers and their family members.

II. Identify the most effective intervention combination that could be delivered for a cost of $364 or less, which is the reimbursement level provided by Medicare for 6 months of intensive behavioral weight loss counseling.

III. Explore the effects of each component on weight loss, vegetable and fruit consumption, percent energy from fat, and physical activity 4 months after the end of the intervention.

IV. Evaluate whether the effects of the intervention components differ by mutation status, previous cancer diagnosis in the index participant, HBOC versus (vs) LS, family environment, and gender of index participant.

V. Pilot test the intervention in MD Anderson's Cancer Prevention Center, to determine the feasibility of providing the intervention components in a clinical setting.

OUTLINE:

Participants are randomized to 1 of 24 conditions, each comprising weight management and health behavior intervention with different combinations of 4 components for 16 weeks. The 4 components are: telephone coaching vs email coaching vs no coaching, text messages vs no text messages, self-monitoring 4-7 days a week vs 1 day per week, and a family team intervention vs none.

TELEPHONE COACHING: Participants receive 1 phone call each week from a coach over 30-45 minutes to discuss diet, physical activity and goal setting.

EMAIL COACHING: Participants receive 1 phone call to discuss the process over 10-15 minutes and then receive 1 email each week for 16 weeks.

NO COACHING: Participants receive 1 phone call the first week over 10-15 minutes to discuss the process.

TEXT MESSAGING: Participants receive 7-12 text messages comprising information about diet and physical activity each week for 16 weeks.

SELF-MONITORING: Participants record their food intake and weight directly into the Fitbit website or application 4-7 days each week or 1 day each week for 16 weeks.

FAMILY TEAM INTERVENTION: Participants (patients and their family members) receive 2 group phone calls and join a Facebook group that is monitored by research staff where they can interact with each other and coaches. The Facebook group includes weekly updates on team progress, weekly family challenges and live online chats with a dietitian and exercise expert.

After completion of study, patients are followed up at 4 and 8 months.

ELIGIBILITY:
Inclusion Criteria:

* HEALTH4Families only: Positive for either HBOC or LS predisposing mutations OR a family member of a mutation carrier (family members do not need to be biological relatives).
* HEALTH4Families only: Index participant ONLY: Must have at least one family member who is eligible and consents to participation.
* Have at least one of the following risk factors:

  * Body mass index (BMI) of 25 or higher
  * < 5 servings of vegetables and fruits per day
  * < 150 minutes per week of moderate intensity activity
  * 75 minutes per week of vigorous intensity activity
* Able to read and write English.
* Have a cellular telephone and are able and willing to send and receive text messages.
* Access to internet via desktop or mobile device.
* Capable of participating in moderate-vigorous unsupervised exercise.
* HEALTH4CPC only: Patient in MD Anderson's Cancer Prevention Center coming in to the clinic for one of the following appointment types: consult and new patient screening appointments
* HEALTH4CPC only: Female.
* HEALTH4CPC only: Lives in the Houston area or surrounding counties (within 150 miles of MD Anderson's main campus).
* HEALTH4CPC only: Has a smartphone.

Exclusion Criteria:

* Unable to walk without crutches, walker, cane, or other assistive device.
* Women who are pregnant or nursing (by self-report).
* Currently receiving radiation therapy or cytotoxic chemotherapy.
* Within 3 months of major surgery.
* Does not live in the United States.
* HEALTH4CPC only: Persons diagnosed with any invasive cancer excluding non-melanoma skin cancer.
* HEALTH4CPC only: Patient at high risk for cancer.
* HEALTH4CPC only: Participated in the HEALTH 4 MD Anderson pilot study (protocol 2014-0230).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2017-01-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Percent weight loss | Baseline to 4 months
  The data from the proposed factorial experiment will be analyzed through analysis of variance (ANOVA) with repeated measures. The outcome variable is the percent weight loss of each participant at 4 months. The fixed covariates include indicator variables for all intervention components. The model includes a random intercept that introduces within-family correlation. The main effect of each intervention component will be tested in an F-test at alpha = 0.0125 level. The pairwise interactions of the intervention components will be studied in an exploratory fashion. The optimal intervention is defined to be the combination of the four components that produces the best percent weight loss result within the resource constraints. Data can also be analyzed jointly in a linear mixed model that includes intervention components and time as fixed effect, family as random intercept and longitudinal correlation between 4 and 8 month data.

SECONDARY OUTCOMES:
Fruit and vegetable consumption | Up to 8 months
  The data from the proposed factorial experiment will be analyzed through ANOVA with repeated measures. The fixed covariates include indicator variables for all intervention components. The model includes a random intercept that introduces within-family correlation. The main effect of each intervention component will be tested in an F-test at alpha = 0.0125 level. Similar ANOVA analysis will be conducted for the 8 month outcome to study whether the intervention effect persists 4 months after the end of the intervention. The 4- and 8-month data can also be analyzed jointly in a linear mixed model that includes intervention components and time as fixed effect, family as random intercept and longitudinal correlation between 4 and 8 month data.
Percent energy from fat | Up to 8 months
  The data from the proposed factorial experiment will be analyzed through ANOVA with repeated measures. The fixed covariates include indicator variables for all intervention components. The model includes a random intercept that introduces within-family correlation. The main effect of each intervention component will be tested in an F-test at alpha = 0.0125 level. Similar ANOVA analysis will be conducted for the 8 month outcome to study whether the intervention effect persists 4 months after the end of the intervention. The 4- and 8-month data can also be analyzed jointly in a linear mixed model that includes intervention components and time as fixed effect, family as random intercept and longitudinal correlation between 4 and 8 month data.
Physical activity | Up to 8 months
  The data from the proposed factorial experiment will be analyzed through ANOVA with repeated measures. The fixed covariates include indicator variables for all intervention components. The model includes a random intercept that introduces within-family correlation. The main effect of each intervention component will be tested in an F-test at alpha = 0.0125 level. Similar ANOVA analysis will be conducted for the 8 month outcome to study whether the intervention effect persists 4 months after the end of the intervention. The 4- and 8-month data can also be analyzed jointly in a linear mixed model that includes intervention components and time as fixed effect, family as random intercept and longitudinal correlation between 4 and 8 month data.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Basen-Engquist, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org